CLINICAL TRIAL: NCT06673563
Title: Development and Evaluation of a Patient-reported Experience Measure (PREM) in Implant Dentistry: an Exploratory Study
Brief Title: A Clinical Study Collecting Patients' Experience During Dental Implant Treatment
Status: Not yet recruiting | Type: Observational
Sponsor: Dr Robert Bowe (Other)
Collaborators: Nobel Biocare (Industry)
Responsible Party: Sponsor-Investigator, Dr Robert Bowe, BA, BDentSc, MFD RCSI, Bowe Dental Clinic
Organization: Bowe Dental Clinic (Other)
Other Study IDs: 2023-1779
Record Dates: First submitted 2024-10-31; First posted 2024-11-05 (Actual); Last update posted 2024-11-05 (Actual); Status verified 2024-11

CONDITIONS: Dental Implant; Dental Restorations; Patient Reported Outcome; Patient Experience

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Single tooth: Patient with the need of a single implant treatment
- Multiple teeth: Patients in need of two or more dental implants
- Full-arch: Patients in need of at least one All-on-4 treatment (with or without additional placed implants)

SUMMARY:
The study will gather data on patient reported experience (PREM) before, during and after dental implant treatment. Patients scheduled in three treatment groups for either single tooth, multiple teeth or full-arch dental rehabilitation are included in the study and will be treated according standard of care. Additionally, they are asked to report their experience based on pre-defined questionnaire assessing patient acceptance of implant treatment in dentistry. Patients will be followed-up until 1-Year post Final Prosthesis Delivery.

This studies primary endpoint is the completion of the PREM questionnaires. The study is not intended to investigate safety and performance of the used medical devices.

ELIGIBILITY:
Inclusion Criteria:

* Subject signed informed consent
* Subject is at least 18 years old at the time of treatment
* Subject presented with the need of dental implant treatment for single tooth, multiple teeth, or full-arch rehabilitation
* Subject with medical and anatomical conditions that are in accordance with the applicable instructions for use (IFU)
* Subject agree to provide information on her/his experience and outcomes before, during and after the treatment
* Subject has a working e-mail address
* Subject has sufficient English language skills for answering the PREM questionnaires

Exclusion Criteria:

* Anatomical conditions discovered during surgery preventing the use of intended implant system
* Subject with history of allergy or adverse reactions to any materials used
* Uncontrolled unstable systemic disease
* Any ongoing application of medication that is interfering with the dental treatment
* Subject is not willing / unable to complete the PREM questionnaires
* Subject that is planning not to return to the investigational site for follow-up visits within study schedule
* Pregnant or lactating women at the time of implant insertion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients in need of a dental implant treatment
Sampling Method: Non-Probability Sample
Enrollment: 99 (Estimated)
Dates: Start 2025-01 (Estimated); Primary Completion 2025-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Patient reported experience at Pre-Treatment, Baseline (Implant Insertion) and Up to 6 months (Final Prosthesis Delivery) | Pre-Treatment, Baseline (Implant Insertion), Up to 6 months (Final Prosthesis Delivery)

SECONDARY OUTCOMES:
Patient reported experience at 1-Year Follow-up | 1-Year Follow-Up
OHIP-14 (summary score and separate questions) | Pre-Treatment, Baseline (Implant Insertion), Up to 6 months (Final Prosthesis Delivery), 1-Year Follow-Up
Patient satisfaction with esthetics and function (VAS) | Pre-Treatment, Baseline (Implant Insertion), Up to 6 months (Final Prosthesis Delivery), 1-Year Follow-Up
Implant survival | Up to 6 months (Final Prosthesis Delivery), 1-Year Follow-Up
Prosthetic survival | 1-Year Follow-Up Visit
Keratinized Mucosa Status | Up to 6 months (Final Prosthesis Delivery), 1-Year Follow-Up
Gingival Index | Up to 6 months (Final Prosthesis Delivery), 1-Year Follow-Up

IPD SHARING:
Plan to Share IPD: No